CLINICAL TRIAL: NCT04067817
Title: Comparison of the Effects of Norepinephrine and Phenylephrine on Tissue Oxygenation and Hemodynamic Stability During an Stroke Volume Variations(SVV) Fluid Guided Therapy in Elderly Undergoing Major Abdominal Surgery
Brief Title: Norepinephrine and Phenylephrine, Which Better for Elderly?
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: poster2016
Record Dates: First submitted 2019-07-20; First posted 2019-08-28 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-07

CONDITIONS: Hypotension
Keywords: Goal-directed Fluid Therapy; norepinephrine; phenylephrine; elderly
MeSH Terms: conditions — Hypotension | interventions — Norepinephrine; Vasoconstrictor Agents; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- norepinephrine (Experimental): Blood pressure is generally maintained at value not less than 80% of baseline during intraoperative period. If the blood pressure is within normal range and SVV is less than 9, patient will be given a continuous infusion of crystalloid solution. However, when blood pressure drops and SVV is greater than 13, a bolus of 200mL colloid will then be quickly administered. If the blood pressure doesn't recover back to normal range within 5 minutes after bolus, norepinephrine will be given through the central venous catheter. If SVV is between 9 and 13, a bolus of crystalloid at 8mL/kg/h will be administered
  Interventions: Drug: norepinephrine
- phenylephrine (Experimental): Blood pressure is generally maintained at value not less than 80% of baseline during intraoperative period. If the blood pressure is within normal range and SVV is less than 9, patient will be given a continuous infusion of crystalloid solution. However, when blood pressure drops and SVV is greater than 13, a bolus of 200mL colloid will then be quickly administered. If the blood pressure doesn't recover back to normal range within 5 minutes after bolus, phenylephrine will be given through the central venous catheter. If SVV is between 9 and 13, a bolus of crystalloid at 8mL/kg/h will be administered.
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: norepinephrine — patient who was received the treatment of norepinephrine
  Other Names: noradrenaline; vasopressor
  Arms: norepinephrine
Drug: Phenylephrine — patient who was received the treatment of phenylephrine
  Other Names: vasopressor
  Arms: phenylephrine

SUMMARY:
this is a prospective, double-blinded and single-center study. this study is based on the Stroke volume variation fluid guided therapy, to compare the effects of norepinephrine and phenylephrine in treating perioperative hypotension, and to find the safest and most effective vasopressor for elderly.

ELIGIBILITY:
Inclusion Criteria:

* radical resection of colorectal or gastric cancers,
* age over 65 years old,
* surgical time longer than 2hours,
* the American Society of Anesthesiologists(ASA) classification of II or III

Exclusion Criteria:

* history of severe cardiovascular diseases,
* history of severe liver and kidney diseases,
* evidence of arrhythmia on EKG,
* use of positive end-expiratory pressure (PEEP) during mechanical ventilation;
* conditions with relative contraindication for arterial catheterization

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-06 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
hemodynamics- (CO)cardiac output | change from patient enters the operating room to end of operation, assessed up to the whole operation
  (CO)cardiac output in Litres per minute. the indicator reflect the patients hemodynamic, which measured by the FloTrac/Vigileo 3.0
Tissue perfusion and oxygenation-(DO2) Oxygen delivery; | change from beginning of operation to end of operation, assessed up to the whole operation
  Blood samples from the radial artery and internal jugular vein were taken at the same time in three time points respectively to measure arterial and venous blood gas, and Measured tissue oxygenation according to Fick equation:DO2(ml/min/m2)=CaO2×10×CI, Arterial oxygen content (CaO2)=Arterial hemoglobin concentration(Hba)×1.36×arterial oxygen saturation(SaO2) + 0.0031×arterial oxygen pressure (PaO2) ;
Tissue perfusion and oxygenation-(VO2)Oxygen consumption; | change from beginning of operation to end of operation, assessed up to the whole operation
  Blood samples from the radial artery and internal jugular vein were taken at the same time in three time points respectively to measure arterial and venous blood gas, and Measured tissue oxygenation according to Fick equation:VO2(ml/min/m2)= (CaO2-CcvO2)×CI×10, Intravenous oxygen content (CcvO2)= Intravenous hemoglobin concentration (Hbv)×1.36×Venous oxygen saturation (ScvO2) + 0.0031×venous oxygen pressure (PcvO2);

CONTACTS AND LOCATIONS:
Overall Officials: xiao z yang, MD,PhD, Study Director — The Second Affiliated Hospital of Dalian Medical University
Locations (1):
- The Second Hospital of Dalian Medical University, Dalian, Liaoning, China